CLINICAL TRIAL: NCT02999503
Title: Nutritional and Environmental Conditions in Attention Deficit Hyperactivity Disorder
Brief Title: Attention Deficit Hyperactivity Disorder: Nutrition and Environment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital El Escorial (Other)
Responsible Party: Principal Investigator, Blumenfeld Olivares JA, Pediatrician, Responsible of Pediatric Endocrinology. Principal Investigator., Hospital El Escorial
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CINUSA1
Record Dates: First submitted 2016-12-01; First posted 2016-12-21 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: ADHD; Lifestyle-Related Condition; Food Habits
Keywords: adhd treatment; nutrition
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Mental Disorders; Feeding Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutritional intervention (Experimental): Patients subject to nutritional education by CINUSA group protocol
  Interventions: Behavioral: Nutritional education
- No intervention (No Intervention): Patients not subject to nutritional education

INTERVENTIONS:
Behavioral: Nutritional education — Nutritional education trough a personal online nutritional consultant
  Arms: Nutritional intervention

SUMMARY:
In this study the investigators aim to investigate the relationship between environmental factors, lifestyle and symptoms of Attention Deficit Hyperactivity Disorder (ADHD). Initially the investigators intend to measure the relationship between nutritional quality, exercise and sleep and ADHD symptoms. And then measure whether a change made in the diet can improve the symptoms of ADHD.

DETAILED DESCRIPTION:
The Attention Deficit Hyperactivity Disorder is a neurobiological chronic disorder, symptomatically evolutionary and of probable genetic transmission that affects between 5 and 10% of the child population.

The current opinion on the etiology of the disorder focuses on a failure in the development of brain circuits in which inhibition and self-control, critical functions to perform any task, gets supported. In addition, there is greater evidence of knowledge of the genetic influence as a major part of the etiology of ADHD. Studies suggest that ADHD is familiar and that genetic influences may contribute to its etiology from moderate to high phenotypic expression. Current studies have identified significant associations with several candidate genes for this disorder, including DAT1, DRD4, DRD5, 5HTT, HTR1B or SNAP25.

Meta-analytical studies are needed to develop a more personalized treatment for ADHD. Other factors associated with ADHD are inadequate lifestyles by parents, especially during the gestation period in the case of the mother. ADHD treatment includes the use of medication and psychosocial and educational support

FOOD, NUTRITION AND ADHD: A NEW PARADIGM OF THERAPY?

Despite the above, with the use of internet many hypotheses have emerged, not yet proven, many in relation to food of patients with ADHD, in which a single focus is exposed as the determinant factor: heavy metals; gluten and dairy; additives; or intake of certain supplements.

The truth is that, neuronal function is strongly influenced by substances in the diet, which are very important for its functioning. Many micronutrients have been evaluated, including mainly vitamins B6, B12, B9, D and E along with some minerals like magnesium, selenium and zinc. Their actions are related to memory, neurotransmitter synthesis and neurological protection.

Multiple studies have found magnesium deficiency in patients with ADHD, as reported in relation to other nutrients. What has also led to study specifically the use of supplementation, in patients with ADHD, with zinc, magnesium, phytochemicals, omega-3 traditional herbs or mixtures of these elements.

OBJECTIVES

* Main objective:

  * Rating, by analysis of results, environmental, nutritional and body composition factors, which may affect the pathogenesis and symptoms of ADHD patients.
* Specific objectives (project sub-lines):

  * Heritage and programming: assessing the hereditary role, as the main factor for the development of ADHD: genetics, nursing, toxic habits in parents and birth characteristics.
  * Diet and physical activity: assessing the role of specific nutrients, eating patterns, exercise, sedentary lifestyle, leisure type and cognitive entertainment, in the development of ADHD.
  * Body Composition: assessing body fat accumulation and muscle mass, aspects involved in the metabolism of people with ADHD.

DESIGN

Cross-sectional study of observational, descriptive and comparative cohort. It consists of volunteer participants, divided into two study groups:

1. cases (ADHD) and
2. controls (healthy, with no ADHD).

For the initial design and protocols main databases have been revised (Scielo, PubMed, ENBASE...).

Development: An observational retrospective cohort study.

Incidental sample: n = 70-100 (approximately 35-50 subjects per group, of the same age range).

Inclusion criteria: both genders, ages 8-16 years.

Intervention trial. A personalized diet for patients will be performed. After completion of the diet, the effect of the intervention on ADHD symptomatology will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Ages 8-16 years
* ADHD proved

Exclusion Criteria:

* Presence of serious or chronic illnesses: leukemia, spinal cord injury, celiac disease, pancreatitis, hepatitis, HIV...

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-05 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Change in Conners | At 3 and 6 months
  Conners conduct questionnaire: attention deficit and disruptive behavior disorders; hyperactivity; and combined type.

SECONDARY OUTCOMES:
Change in sleep | At 3 and 6 months
  Markers related to sleep: adapted Short Form Health Survey-36 for sleep quality.
Change in exercise markers | At 3 and 6 months
  Markers related to activity: Ipad-Minnesota questionnaire for physical activity.
Change in Anthropometry I | At 3 and 6 months
  Arm circumference and triceps skinfold, muscle area and arm fat area using the manual for evaluation of body composition in humans of the Spanish population.
Change in Anthropometry II | At 3 and 6 months
  BMI, calculated using height and weight.
Change in Anthropometry III | At 3 and 6 months
  % total body fat,% visceral fat,% muscle. Measured by electrical bioimpedance, apparatus for medical use which analyzes the opposition of a biological tissue (fat) to the passage of an electric current through it. It is a noninvasive, painless study based on the application of an electrical current through the body and the record of physical parameters that depend on body's water content. The investigators will use a M230 InBody bioimpedance, multi-frequency (20 to 100 Hz), tetra-pole or similar.
Change in Anthropometry IV | At 3 and 6 months
  Arm circumference and triceps skinfold, muscle area and arm fat area using the manual for evaluation of body composition in humans of the Spanish population.
Change in nutritional habits | At 3 and 6 months
  Kidmed ( mediterranean diet adherence) questionnaire at baseline, 3 and 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Javier Andres Blumenfeld Olivares, MD, Principal Investigator — Hospital El Escoral
Locations (1):
- Hospital EL Escorial, El Escorial, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gillies D, Leach MJ, Perez Algorta G. Polyunsaturated fatty acids (PUFA) for attention deficit hyperactivity disorder (ADHD) in children and adolescents. Cochrane Database Syst Rev. 2023 Apr 14;4(4):CD007986. doi: 10.1002/14651858.CD007986.pub3. PMID 37058600